CLINICAL TRIAL: NCT07089446
Title: Combination of Platelets Rich Plasma and Hyaluronic is an Effective Tool for Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Karachi (Other)
Responsible Party: Principal Investigator, Dr Ranjeet Kumar, Principal investigator, University of Karachi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCH-IRB-2022-05
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthristis
Keywords: Hyaluronic acid; osteoarthritis; pain; disability
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Participants were randomly divided into three groups. Twenty cases (Group A) were injected with HA, 20 (Group B) had PRP, and the remaining 20 (Group C) received a combination of HA and PRP
Who Masked: Outcomes Assessor
Masking Description: Single blinded study, only the assessor was kept blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Hyaluronic acid
  Interventions: Drug: Hyaluronic Acid (HA)
- Group B (Active Comparator): platelet rich plasma
  Interventions: Drug: Platelet Rich Plasma
- Group C (Other): Hyaluronic acid and platelet rich plasma
  Interventions: Drug: Hyaluronic Acid (HA) and Platelet rich plasma

INTERVENTIONS:
Drug: Hyaluronic Acid (HA) — Hyaluronic Acid
  Arms: Group A
Drug: Platelet Rich Plasma — Platelet rich plasma
  Arms: Group B
Drug: Hyaluronic Acid (HA) and Platelet rich plasma — Hyaluronic Acid and Platelet rich plasma
  Arms: Group C

SUMMARY:
The purpose of the study is to determine the effects of HA, PRP and the combination of HA and PRP in reducing pain and improving functional disability in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
To determine the effects of combination of platelet rich plasma (PRP) and hyaluronic acid and the PRP or HA alone in reducing pain and increasing range of motion among individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* grade II-III according to the Kellgren-Lawrence classification),
* pain or functional limitations in patients' activity of daily living before the treatment,
* age between 40 and 70 years of age, and the absence of clinical or imaging signs of articular instability.

Exclusion Criteria:

* includes known hypersensitivity to hyaluronic acid,
* pregnancy and lactation, a BMI greater than 40 kg/m2,
* chronic administration of anticoagulant drugs or a history of coagulopathies,
* neoplastic lesions, and knee or kidney failures

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | Recorded before the treatment and repeated within 3 and 6 months after the treatment.
  It is a straight line, 100 millimeters long line, one end of the line means "not at all" or "none" and the other end means "the worst possible" or "extremely".

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Recorded before the treatment and repeated within 3 and 6 months after the treatment.
  It s a questionnaire used to assess pain, stiffness, and physical function in individuals with osteoarthritis, particularly of the knee. It is a self-administered, multidimensional tool that evaluates these three dimensions through a series of questions, typically on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Basit Ansari, PhD, Study Chair — University of Karachi; Ranjeet Kumar, MBBS, FCPS, Principal Investigator — University of Karachi; Aftab Ahmed Mirza Baig, PhD, Study Director — IQRA University
Locations (1):
- South City Hospital, Karachi, Sindh, Pakistan